CLINICAL TRIAL: NCT06872047
Title: Exploring the Knowledge, Attitudes, Behaviors and Perceived Barriers of Hepatologists Towards Non-invasive Hepatocellular Carcinoma Prediction Models in Hepatitis C Patients Who Achieved Sustained Virological Response Following Direct Acting Antivirals Therapy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aalaa Mahmoud Younis, residant doctor, Assiut University
Other Study IDs: KAP Hepatologists HCC HCV pt
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Non-invasive Hepatocellular Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group A: hepatologists dealing with patients with hepatocellular carcinoma (HCC) in patients with chronic hepatitis C (HCV) who achieved sustained virological response (SVR) after direct-acting antiviral (DAA) therapy.

SUMMARY:
This study aims to assess the knowledge, attitudes, and behaviors (KAB) of hepatologists regarding different models used to predict hepatocellular carcinoma (HCC) in patients with chronic hepatitis C (HCV) who achieved sustained virological response (SVR) after direct-acting antiviral (DAA) therapy. The study will use a structured questionnaire targeting hepatologists globally to evaluate their familiarity with, confidence in, and clinical application of various predictive models. The primary outcome is the proportion of hepatologists who incorporate prediction models in clinical practice, while secondary outcomes include the level of knowledge about different models, perceived reliability, and barriers to their implementation the aim of the study 1) To evaluate the level of knowledge among hepatologists regarding existing HCC prediction models for post-SVR HCV patients.

2) To assess hepatologists' attitudes toward the utility, reliability, and clinical value of these models.

3) To identify the extent to which hepatologists incorporate predictive models into their clinical decision-making.

4) To determine perceived barriers to the adoption of these models in clinical practice.

5) To explore the factors associated with poor adoption of these predictive models.

ELIGIBILITY:
Inclusion Criteria:

* Hepatologists with at least one year of experience in managing HCV patients

Exclusion Criteria:

* Non-hepatologists, general practitioners, or respondents who submit incomplete surveys

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Practicing hepatologists involved in the management of HCV patients.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
percentage of hepatologists who use HCC prediction models in clinical practice. | baseline
  The percentage of hepatologists who use HCC prediction models in clinical practice.